CLINICAL TRIAL: NCT02972632
Title: An Open-Label, Single-Arm, Multicenter, Prospective, Phase 4, Interventional, Flexible Dose Study to Evaluate the Effectiveness of Vortioxetine on Goal Achievement After a Change in Antidepressant Medication for the Treatment of Subjects With Major Depressive Disorder
Brief Title: Goal Achievement After a Change to Vortioxetine in Adults With Major Depressive Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Vortioxetine-4003; U1111-1185-6902 (Other: WHO)
Record Dates: First submitted 2016-11-21; First posted 2016-11-23 (Estimated); Results first posted 2019-07-11 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-06

CONDITIONS: Major Depressive Disorder
Keywords: Drug Therapy
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Vortioxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vortioxetine 10-20 mg (Experimental): Vortioxetine 10 mg, tablets, orally, once daily followed by a dose adjustment to a maximum of 20 mg, tablets, orally, once daily up to 12 weeks. The dose may be decreased by 5 mg based on participant's response and tolerability as judged by the investigator.
  Interventions: Drug: Vortioxetine

INTERVENTIONS:
Drug: Vortioxetine — Vortioxetine tablet
  Other Names: LuAA21004

SUMMARY:
The purpose of this study is to determine the effectiveness of treatment with vortioxetine on participant goal achievement after a change in antidepressant medication for the treatment of major depressive disorder (MDD).

DETAILED DESCRIPTION:
The drug being tested in this study is called Vortioxetine. Vortioxetine is being tested to treat depression in people who have major depressive disorder. This study will look at effectiveness of treatment with vortioxetine in participant's goal achievement for the treatment of major depressive disorder.

The study enrolled 123 patients. Participants will receive:

• Vortioxetine 10 to 20 mg

All participants will be asked to take one tablet at the same time each day throughout the study. The participants will receive a starting dose of 10 mg. The dose may be up-titrated to 20 mg. The dose may then be decreased by 5 mg based on participant's response and tolerability to higher dose as judged by the Investigator.

This multi-center trial will be conducted in Unites States. The overall time to participate in this study is 19 weeks. Participants will make multiple visits to the clinic and will be contacted by telephone for 4 weeks after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Is suffering from Major Depressive Disorder (MDD) as the primary psychiatric diagnosis.
2. Has been or is currently being treated with an approved antidepressant (monotherapy) for 6 weeks or longer at an adequate therapeutic dose. Participants currently on an antidepressant at Screening will be discontinued in a manner that is consistent with labeling recommendations and conventional medical practice.
3. The antidepressant treatment must be on-going at time of Screening or have been discontinued within the 6 weeks prior to Screening.
4. Is considered appropriate for a change in antidepressant medication based on Investigator judgment in collaboration with the participant.
5. Has scores on Patient Health Questionnaire (PHQ-9) ≥5 and Clinical Global Impression Scale Severity (CGI-S ≥4).

Exclusion Criteria:

1. Has discontinued prior antidepressant treatment greater than 6 weeks from Screening.
2. Is considered to be at imminent risk for hospitalization due to severe depression in the opinion of the investigator. Recent hospitalization due to MDD within 3 months prior to Screening is exclusionary also.
3. Has a significant risk of suicide according to the Investigator's clinical judgment or has made an actual suicide attempt in the previous 6 months prior to Screening or scores "yes" on items 4 or 5 in the past 6 months on the Suicidal Ideation section of the Columbia Suicide Severity Rating Scale (C-SSRS).
4. Is considered to be treatment resistant, defined as participants with MDD who have not responded to 2 or more separate different antidepressant monotherapy trials of adequate dose and duration (6 weeks or longer) in their current episode. History of only responding to combination or augmentation therapy in previous major depressive episode (MDEs) is also considered evidence of treatment resistant depression.
5. Has 1 or more of the following:

   1. Current or history of: manic or hypomanic episode, schizophrenia or any other psychotic disorder, including schizoaffective disorder, major depression with psychotic features, bipolar depression with psychotic features, obsessive compulsive disorder, mental retardation, organic mental disorders, or mental disorders due to a general medical condition as defined in Diagnostic and Statistical Manual of Mental Disorders (DSM-5) as determined by the investigator.
   2. Current diagnosis or history of alcohol or other substance abuse or dependence (excluding nicotine or caffeine). The participants must have a negative urine drug screen (UDS) at Screening and Baseline, this includes benzodiazepines and opiates (including oxycodone) for which there is no prescription.
   3. Presence or history of a clinically significant neurological disorder (including epilepsy) as determined by the investigator.
   4. Neurodegenerative disorder (Alzheimer disease, Parkinson disease, multiple sclerosis, Huntington disease, etc).
6. Has a known history of acute narrow-angle glaucoma or is at risk of acute narrow-angle glaucoma.
7. Has a known unstable thyroid disorder or a thyroid-stimulating hormone value outside the normal range based on medical history that is deemed clinically significant by the investigator.
8. Has active hepatitis B or a known history of hepatitis C virus.
9. Has a known history of human immunodeficiency virus infection.
10. Has a history of gastric bypass.
11. Has previously or is currently participating in this study or another vortioxetine or LuAA21004 study.
12. Is receiving or who have started receiving formal cognitive or behavioral therapy, systematic psychotherapy within 30 days from screening or plan to initiate such therapy during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2016-12-22 (Actual); Primary Completion 2018-02-06 (Actual); Study Completion 2018-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (25):
- United States (25):
  - ATP Clinical Research, Inc., Costa Mesa, California
  - ProScience Research Group, Culver City, California
  - Behavioral Research Specialists, LLC, Glendale, California
  - Pacific Research Partners, Oakland, California
  - Excell Research, Oceanside, California
  - Anderson Clinical Research, Redlands, California
  - University Medical Group, Upland, California
  - MCB Clinical Research Centers, LLC, Colorado Springs, Colorado
  - Suncoast Clinical Research Inc., New Port Richey, Florida
  - Behavioral Clinical Research , Inc, North Miami, Florida
  - Compass Research Main, Orlando, Florida
  - University of South Florida, Tampa, Florida
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Baber Research Group, Naperville, Illinois
  - Deaconess Clinic, Evansville, Indiana
  - Novex Clinical Research, LLC, New Bedford, Massachusetts
  - Coastal Research Associates, Inc., South Weymouth, Massachusetts
  - University of Michigan, Ann Arbor, Ann Arbor, Michigan
  - Columbia University Medical Center, New York, New York
  - Dayton Clinical Research, Dayton, Ohio
  - Green & Seidner Family Practice Associates, Lansdale, Pennsylvania
  - Relaro Medical Trials, Dallas, Texas
  - Red Oak Psychiatry Associates, PA, Houston, Texas
  - Radiant Research, Inc., San Antonio, Texas
  - Family Psychiatry of The Woodlands, The Woodlands, Texas

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available after applicable marketing approvals and commercial availability have been received, an opportunity for the primary publication of the research has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com/Approach for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

REFERENCES:
- [Derived] McCue M, Sarkey S, Eramo A, Francois C, Parikh SV. Using the Goal Attainment Scale adapted for depression to better understand treatment outcomes in patients with major depressive disorder switching to vortioxetine: a phase 4, single-arm, open-label, multicenter study. BMC Psychiatry. 2021 Dec 11;21(1):622. doi: 10.1186/s12888-021-03608-1. PMID 34895181

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 23 investigative sites in United States from 22 December 2016 to 06 February 2018.
Pre-assignment Details: Participants with a diagnosis of major depressive disorder were enrolled to receive vortioxetine with a starting dose of 10 mg for 12 weeks. Dose was increased or decreased as per investigator's discretion.
Groups:
- Vortioxetine: Vortioxetine 10 mg, tablets, orally, once daily up to 12 weeks. Dose was increased or decreased as per investigator's discretion.
Period: Overall Study
Arm/Group | Vortioxetine
Started | 123
Safety Analysis Set (All participants who received at least one dose study drug.) | 122
Completed | 106
Not Completed | 17
Not completed — Pretreatment Event/Adverse Event | 3
Not completed — Lost to Follow-up | 4
Not completed — Voluntary Withdrawal | 10

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who were enrolled and received at least one dose of study drug.
Arm/Group | Vortioxetine
Number analyzed (Participants) | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (12.22)
Age, Customized [Count of Participants; unit: Participants]
  <= 55 Years | 95
  > 55 Years | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101
  Male | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 28
  Not Hispanic or Latino | 94
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 5
  Black or African American | 28
  Native Hawaiian or Other Pacific Islander | 1
  White | 83
  Multiracial | 3
  Unknown | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 122
Height [Mean (Standard Deviation); unit: cm] | 164.5 (10.43)
Weight [Mean (Standard Deviation); unit: kg] | 91.59 (23.118)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index = weight (kg)/[height (m)^2]
  kg/m^2 | 34.13 (9.666)
Smoking Classification [Count of Participants; unit: Participants]
  Never smoked | 75
  Current smoker | 23
  Ex-smoker | 24

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved Goal Attainment Scale (GAS) Score of ≥50 at Week 12
Description: GAS is a tool to measure progress each participant has towards achieving their individualized goals. The standardized scoring was applied for statistical analysis. A semi-structured interview was conducted with each participant to conduct goal-setting at the outset of study. Another evaluation took place at end of study (EOS) visit to determine the level of progress at that time. The score for each goal ranged from -2 (much worse) to +2 (much better). GAS yielded a norm-based score standardized to a mean of 50 with a standard deviation (SD) of 10. Higher score indicates composite of 3 goals (50 or above) as response.
Time Frame: Week 12
Population: Full analysis set (FAS) included all participants who were enrolled in the treatment period and received at least one dose of the study drug and completed at least one GAS assessment postbaseline. Overall number of participants analyzed is the number of participants with evaluable data at the given time-point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vortioxetine
Number analyzed (Participants) | 109
percentage of participants | 57.8 [48.5 to 67.1]

2. Secondary Outcome: Change From Baseline in Total Goal Attainment Scale Score at Weeks 6 and 12
Description: GAS is a tool to measure progress each participant has towards achieving their individualized goals. The standardized scoring was applied for statistical analysis. A semi-structured interview was conducted with each participant to conduct goal-setting at outset of study. Another evaluation took place at EOS visit to determine level of progress at that time. The score for each goal ranged from -2 (much worse) to +2 (much better). GAS yielded a norm-based score standardized to a mean of 50 with SD of 10. The total score ranges between 22.6 and 77.4. A positive change from baseline in the composite of 3 goals (50 or above) indicates response.
Time Frame: Baseline and Weeks 6 and 12
Population: FAS included all participants who were enrolled in the treatment period and received at least one dose of the study drug and completed at least one GAS assessment postbaseline. Number analyzed is the number of participants with evaluable data at the given time-point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vortioxetine
Number analyzed (Participants) | 116
score on a scale
  Baseline | 23.57 (0.073)
  Change at Week 6: number analyzed (Participants) | 110
  Change at Week 6 | 18.21 (11.470)
  Change at Week 12: number analyzed (Participants) | 109
  Change at Week 12 | 26.94 (13.582)
Statistical Analysis 1: Comparison: Vortioxetine; Change at Week 6 relative to baseline; Test type: Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Vortioxetine; Change at Week 12 relative to baseline; Test type: Other; p < 0.001, t-test, 2 sided

3. Secondary Outcome: Change From Baseline in Patient Health Questionnaire (PHQ-9) Score at Weeks 6 and 12
Description: PHQ-9 is a well-established participant reported outcome tool for assessment of change in depressive symptoms and is a sensitive measure of depression severity. The PHQ-9 consists of a 9-item scale originally developed for primary care settings, with 1 item corresponding to each of the 9 made symptom criteria for depression in diagnostic and statistical manual of mental disorders (DSM), asking if they have bothered the participant over the last 2 weeks. Each question is rated on a scale from 0 (not at all) to 3 (nearly every day). If any problems are answered 1 or higher, a final question on how difficult those problems made it to do work, take care of things at home, or get along with other people is completed, rated from not difficult at all to extremely difficult. The 9 questions are summed to a total score ranging from 0 to 27 with higher scores reflecting greater severity. A positive change from baseline indicates severe condition.
Time Frame: Baseline and Weeks 6 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vortioxetine
Number analyzed (Participants) | 116
score on a scale
  Baseline: number analyzed (Participants) | 110
  Baseline | 15.7 (4.79)
  Change at Week 6: number analyzed (Participants) | 103
  Change at Week 6 | -6.5 (6.15)
  Change at Week 12: number analyzed (Participants) | 106
  Change at Week 12 | -8.4 (6.22)
Statistical Analysis 1: Comparison: Vortioxetine; Change at Week 6 relative to baseline; Test type: Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Vortioxetine; Change at Week 12 relative to baseline; Test type: Other; p < 0.001, t-test, 2 sided

4. Secondary Outcome: Change From Baseline in Perceived Deficits Questionnaire-Depression (PDQ-D) at Weeks 6 and 12
Description: The PDQ-D is a 20-item, patient-reported questionnaire with a 7-day recall period. Scores for four subscales. All 20 items use the same 5-point ordinal categorical response scale to reflect the frequency of experiencing a specific cognitive problem in the past 7 days. Scores for each of the four measured subscales are calculated by assigning a value of 0 ("never in the past 7 days"), 1 ("rarely - once or twice"), 2 ("sometimes - 3-5 times"), 3 ("often - about once a day"), or 4 ("very often - more than once a day") to each item, then summing the five items of that subscale, to produce a score ranging from 0 to 20. A total global score for overall cognitive dysfunction (range 0-80) is calculated by summing the four subscale scores. Higher scores for each subscale and for the total score indicate greater perceived cognitive dysfunction. A negative change from Baseline indicates improvement.
Time Frame: Baseline and Weeks 6 and 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vortioxetine
Number analyzed (Participants) | 116
score on a scale
  Baseline: number analyzed (Participants) | 110
  Baseline | 40.5 (14.87)
  Change at Week 6: number analyzed (Participants) | 104
  Change at Week 6 | -14.8 (13.70)
  Change at Week 12: number analyzed (Participants) | 106
  Change at Week 12 | -18.0 (16.92)
Statistical Analysis 1: Comparison: Vortioxetine; Change at Week 6 relative to baseline; Test type: Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Vortioxetine; Change at Week 12 relative to baseline; Test type: Other; p < 0.001, t-test, 2 sided

5. Secondary Outcome: Change From Baseline in Quality of Life Enjoyment and Satisfaction Scale (Q-LES-Q) Total Score at Week 12
Description: Q-LES-Q is a scale designed to allow researchers to assess the degree of a participant's quality of life in various areas of daily living. There is not a "Total Score" per se for the Q-LES-Q. The scale is divided into domains. Ninety-one of the 93 items are assembled into 8 categories: physical health/activities, feelings, work, household duties, school/course work, leisure time activities, social relations, and general activities. Items are scored on a 5 point scale, from 1 (not at all or never) to 5 (frequently or all the time), to indicate the degree of enjoyment or satisfaction experienced by domain. Raw summary scores are expressed as a percentage of the maximum possible score within a given domain to facilitate comparisons across areas of functioning. The total score is based on the Overall Life Satisfaction question in General Activities and ranges from 1 to 5. A positive change from baseline indicates greater enjoyment/satisfaction.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vortioxetine
Number analyzed (Participants) | 116
score on a scale
  Baseline: number analyzed (Participants) | 115
  Baseline | 2.487 (0.8822)
  Change at Week 12: number analyzed (Participants) | 109
  Change at Week 12 | 1.128 (1.1871)
Statistical Analysis 1: Comparison: Vortioxetine; Change at Week 12 relative to baseline; Test type: Other; p < 0.001, t-test, 2 sided

6. Secondary Outcome: Change From Baseline in 5-Item World Health Organization Well-being Index (WHO-5) Score at Week 12
Description: WHO-5 is a short, self-administered questionnaire covering 5 positively worded items, related to positive mood (good spirits, relaxation), vitality (being active and waking up fresh and rested), and general interests (being interested in things). Each of the five items is rated from 0 (= not present) to 5 (= constantly present). Scores are summated, with raw score ranging from 0 to 25, with higher score meaning better well-being. A positive change from baseline indicates improvement.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vortioxetine
Number analyzed (Participants) | 116
score on a scale
  Baseline: number analyzed (Participants) | 115
  Baseline | 5.6 (3.48)
  Change at Week 12: number analyzed (Participants) | 109
  Change at Week 12 | 7.2 (6.59)
Statistical Analysis 1: Comparison: Vortioxetine; Change at Week 12 relative to baseline; Test type: Other; p < 0.001, t-test, 2 sided

7. Secondary Outcome: Change From Baseline in Clinical Global Impression Scale Severity (CGI-S) at Week 12
Description: CGI-S is a clinician rated scale designed to assess global severity of illness and change in the clinical condition over time. The CGI-S provides the clinician's impression of the participant's state of mental illness. The clinician uses his or her clinical experience of this participant population to rate the severity of the participant's mental illness on a 7-point scale ranging from 1 (normal-not at all ill) to 7 (among the most extremely ill participants). Higher scores indicate greater severity of illness. A negative change from baseline indicates improvement.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vortioxetine
Number analyzed (Participants) | 116
score on a scale
  Baseline: number analyzed (Participants) | 114
  Baseline | 4.4 (0.50)
  Change at Week 12: number analyzed (Participants) | 110
  Change at Week 12 | -1.6 (1.10)
Statistical Analysis 1: Comparison: Vortioxetine; Change at Week 12 relative to baseline; Test type: Other; p < 0.001, t-test, 2 sided

8. Secondary Outcome: Clinical Global Impression Scale-Improvement (CGI-I) Score at Week 12
Description: CGI-I assesses the participant's improvement (or worsening). The clinician assessed participant's condition on a 7-point scale ranging from 1 (very much improved) to 7 (very much worse). Higher scores indicated greater severity of illness.
Time Frame: Week 12
Population: FAS included all participants who were enrolled in the treatment period and received at least one dose of the study drug and completed at least one GAS assessment postbaseline. Overall number of participants analyzed is the number of participants with evaluable data at the given time-point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vortioxetine
Number analyzed (Participants) | 111
score on a scale | 2.2 (1.05)

ADVERSE EVENTS:
Time Frame: Baseline up to Day 113
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Safety analysis set included all participants who were enrolled and received at least one dose of study drug.
Arm/Group | Vortioxetine
All-Cause Mortality (participants affected / at risk) | 0/122
Serious Adverse Events (participants affected / at risk) | 1/122
Other Adverse Events (participants affected / at risk) | 46/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vortioxetine (N=122)
Depression (Psychiatric disorders) | 1
Suicidal Ideation (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vortioxetine (N=122)
Nausea (Gastrointestinal disorders) | 26
Constipation (Gastrointestinal disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 7
Headache (Nervous system disorders) | 11
Anxiety (Psychiatric disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-02-15): https://cdn.clinicaltrials.gov/large-docs/32/NCT02972632/SAP_000.pdf
  • Study Protocol (2017-08-18): https://cdn.clinicaltrials.gov/large-docs/32/NCT02972632/Prot_001.pdf